CLINICAL TRIAL: NCT02663362
Title: Development and Validation of Multi-nuclear Magnetic Resonance Imaging and Spectroscopy for Whole Body Human Applications
Acronym: MRS VALIDATION
Status: Recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMD FH 306624
Record Dates: First submitted 2016-01-14; First posted 2016-01-26 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Human Body Composition; Human Body Function
Keywords: magnetic resonance imaging; magnetic resonance spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: To evaluate the reproducibility of acquiring multi-nuclear data on a new 3T Philips Magnet — Outside standard MR instrumentation there will be no interventions.

SUMMARY:
The purpose of this study is to develop and refine the techniques for using magnetic resonance imaging and magnetic resonance spectroscopy to understand the composition and function of the human body

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 12 - 89
* Healthy (self assessed)
* Weight under 350lbs
* Able to walk 50 yards without stopping
* Able to travel to hospital for study visits
* Able to follow a 3-step command
* Able to remain in Magnetic Resonance (MR) scanner for up to 2 hours

Exclusion Criteria:

* Have internal metal medical devices, including cardiac pacemakers, aortic or cerebral aneurysm clips, artificial heart valves, ferromagnetic implants, shrapnel, wire sutures, joint replacements, bone or joint pins/rods/screws, metal fragments in your eye, or non-removable jewelry such as rings.
* Are unwilling or unable to complete the imaging procedures for the duration of the MRI scan due to claustrophobia or other reason.
* Serious mental illness that might preclude subject's ability to comply with study treatment
* Life expectancy of less than 1 year
* Are pregnant or plan on becoming pregnant in the next 8 weeks.

Ages: 12 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A healthy individual, who is willing and able to undergo MR imaging and spectroscopy for up to two hours at a time
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-02; Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Whole body fat quantification | 1 hour

SECONDARY OUTCOMES:
Fat Microstructure | 1 hour
  A high resolution image of the structure of fat tissue.

OTHER OUTCOMES:
Flow high resolution imaging | 1 hour
  Image of the movement of fluids in the area being imaged.
Intramyocellular fat quantification | 45 minutes
  Use to determine the amount and types of fat inside muscle and liver.
Intrahepatic fat quantification | 45 minutes
  A measure of the amount of fat in the liver.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Cornnell, PhD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tyler DJ, Hudsmith LE, Clarke K, Neubauer S, Robson MD. A comparison of cardiac (31)P MRS at 1.5 and 3 T. NMR Biomed. 2008 Oct;21(8):793-8. doi: 10.1002/nbm.1255. PMID 18512846
- [Background] Muller HP, Raudies F, Unrath A, Neumann H, Ludolph AC, Kassubek J. Quantification of human body fat tissue percentage by MRI. NMR Biomed. 2011 Jan;24(1):17-24. doi: 10.1002/nbm.1549. PMID 20672389
- [Background] Price RR, Allison J, Massoth RJ, Clarke GD, Drost DJ; NMR Task Group #8. Practical aspects of functional MRI (NMR Task Group #8). Med Phys. 2002 Aug;29(8):1892-912. doi: 10.1118/1.1494990. PMID 12201436
- [Background] Noseworthy MD, Bulte DP, Alfonsi J. BOLD magnetic resonance imaging of skeletal muscle. Semin Musculoskelet Radiol. 2003 Dec;7(4):307-15. doi: 10.1055/s-2004-815678. PMID 14735429
- [Background] Lebon V, Dufour S, Petersen KF, Ren J, Jucker BM, Slezak LA, Cline GW, Rothman DL, Shulman GI. Effect of triiodothyronine on mitochondrial energy coupling in human skeletal muscle. J Clin Invest. 2001 Sep;108(5):733-7. doi: 10.1172/JCI11775. PMID 11544279
- [Background] Roser W, Beckmann N, Wiesmann U, Seelig J. Absolute quantification of the hepatic glycogen content in a patient with glycogen storage disease by 13C magnetic resonance spectroscopy. Magn Reson Imaging. 1996;14(10):1217-20. doi: 10.1016/s0730-725x(96)00243-3. PMID 9065913
- [Background] Beckmann N, Fried R, Turkalj I, Seelig J, Keller U, Stalder G. Noninvasive observation of hepatic glycogen formation in man by 13C MRS after oral and intravenous glucose administration. Magn Reson Med. 1993 May;29(5):583-90. doi: 10.1002/mrm.1910290502. PMID 8505893
- [Background] van der Meer RW, Doornbos J, Kozerke S, Schar M, Bax JJ, Hammer S, Smit JW, Romijn JA, Diamant M, Rijzewijk LJ, de Roos A, Lamb HJ. Metabolic imaging of myocardial triglyceride content: reproducibility of 1H MR spectroscopy with respiratory navigator gating in volunteers. Radiology. 2007 Oct;245(1):251-7. doi: 10.1148/radiol.2451061904. PMID 17885193
- [Background] Schar M, Kozerke S, Boesiger P. Navigator gating and volume tracking for double-triggered cardiac proton spectroscopy at 3 Tesla. Magn Reson Med. 2004 Jun;51(6):1091-5. doi: 10.1002/mrm.20123. PMID 15170826
- [Background] Hudsmith LE, Tyler DJ, Emmanuel Y, Petersen SE, Francis JM, Watkins H, Clarke K, Robson MD, Neubauer S. (31)P cardiac magnetic resonance spectroscopy during leg exercise at 3 Tesla. Int J Cardiovasc Imaging. 2009 Dec;25(8):819-26. doi: 10.1007/s10554-009-9492-8. Epub 2009 Aug 21. PMID 19697152
- [Background] Shen W, Mao X, Wang Z, Punyanitya M, Heymsfield SB, Shungu DC. Measurement of intramyocellular lipid levels with 2-D magnetic resonance spectroscopic imaging at 1.5 T. Acta Diabetol. 2003 Oct;40 Suppl 1(Suppl 1):S51-4. doi: 10.1007/s00592-003-0026-x. PMID 14618433
- [Background] Shen W, Mao X, Wolper C, Heshka S, Dashnaw S, Hirsch J, Heymsfield SB, Shungu DC. Reproducibility of single- and multi-voxel 1H MRS measurements of intramyocellular lipid in overweight and lean subjects under conditions of controlled dietary calorie and fat intake. NMR Biomed. 2008 Jun;21(5):498-506. doi: 10.1002/nbm.1218. PMID 17955571
- [Background] Larson-Meyer DE, Newcomer BR, Hunter GR. Influence of endurance running and recovery diet on intramyocellular lipid content in women: a 1H NMR study. Am J Physiol Endocrinol Metab. 2002 Jan;282(1):E95-E106. doi: 10.1152/ajpendo.2002.282.1.E95. PMID 11739089
- [Background] Larson-Meyer DE, Smith SR, Heilbronn LK, Kelley DE, Ravussin E, Newcomer BR; Look AHEAD Adipose Research Group. Muscle-associated triglyceride measured by computed tomography and magnetic resonance spectroscopy. Obesity (Silver Spring). 2006 Jan;14(1):73-87. doi: 10.1038/oby.2006.10. PMID 16493125
- [Background] Positano V, Gastaldelli A, Sironi AM, Santarelli MF, Lombardi M, Landini L. An accurate and robust method for unsupervised assessment of abdominal fat by MRI. J Magn Reson Imaging. 2004 Oct;20(4):684-9. doi: 10.1002/jmri.20167. PMID 15390229
- [Background] Smith SR, Lovejoy JC, Greenway F, Ryan D, deJonge L, de la Bretonne J, Volafova J, Bray GA. Contributions of total body fat, abdominal subcutaneous adipose tissue compartments, and visceral adipose tissue to the metabolic complications of obesity. Metabolism. 2001 Apr;50(4):425-35. doi: 10.1053/meta.2001.21693. PMID 11288037
- [Background] Larson-Meyer DE, Newcomer BR, Hunter GR, Joanisse DR, Weinsier RL, Bamman MM. Relation between in vivo and in vitro measurements of skeletal muscle oxidative metabolism. Muscle Nerve. 2001 Dec;24(12):1665-76. doi: 10.1002/mus.1202. PMID 11745976
- [Background] Larson-Meyer DE, Newcomer BR, Hunter GR, Hetherington HP, Weinsier RL. 31P MRS measurement of mitochondrial function in skeletal muscle: reliability, force-level sensitivity and relation to whole body maximal oxygen uptake. NMR Biomed. 2000 Jan;13(1):14-27. doi: 10.1002/(sici)1099-1492(200002)13:13.0.co;2-0. PMID 10668050
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org